CLINICAL TRIAL: NCT00840684
Title: A PHASE I-II MULTICENTER STUDY OF THE CLORETAZINE-DAUNORUBICIN-ARACYTINE COMBINATION FOR THE TREATMENT OF ACUTE MYELOID LEUKEMIA (AML) WITH UNFAVORABLE CYTOGENETICS
Brief Title: Laromustine, Daunorubicin, and Cytarabine in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000634230; IPC-LAM-HR; IPC-2006-007; INCA-RECF0902; EUDRACT-2007-001082-15
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — Amsacrine; Busulfan; Cytarabine; Daunorubicin; laromustine; Melphalan; Mitoxantrone

INTERVENTIONS:
Drug: amsacrine
Drug: busulfan
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: laromustine
Drug: melphalan
Drug: mitoxantrone hydrochloride
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: autologous hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as laromustine, daunorubicin, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of laromustine when given together with daunorubicin and cytarabine in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the dose of laromustine that can be combined with daunorubicin hydrochloride and cytarabine in patients with previously untreated acute myeloid leukemia with unfavorable cytogenetics. (Phase I)
* To determine the complete remission rate of this regimen as induction therapy. (Phase II)

Secondary

* To determine the complete response rate.
* To determine the safety profile of this regimen.
* To determine the overall and relapse-free survival.
* To evaluate the prognostic value of the molecular markers FLT3, duplications of MLL, and Evi-1.

OUTLINE: This is a multicenter, phase I dose-escalation study of laromustine followed by a phase II study.

* Induction treatment: Patients receive laromustine IV on day 4, daunorubicin hydrochloride IV on days 1-3, and cytarabine IV continuously on days 1-7. Patients not attaining complete remission (CR) after first induction receive a second induction treatment comprising daunorubicin hydrochloride IV on days 1-3 and cytarabine IV twice daily on days 1-4. Patients in CR after 1 or 2 induction treatments proceed to consolidation treatment.
* Consolidation treatment: Patients receive mini-consolidation treatment comprising amsacrine on day 1 and cytarabine IV twice daily on days 1-5 followed by 2 courses of continuing consolidation treatment comprising mitoxantrone hydrochloride on days 1 and 2 and cytarabine IV over 12 hours on days 1-5.
* Allogeneic or autologous stem cell transplantation: Patients receive busulfan four times daily for 4 days and melphalan followed by allogeneic or autologous stem cell transplantation.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)

  * Untreated disease
  * No promyelocytic AML
* Unfavorable prognosis, defined as at least one of the following:

  * Cytogenetic abnormalities including -5/5q-, -7/7q-, 3q, 11q23, t(6;9), and complex abnormalities (≥ 3 clonal abnormalities), excluding t(9;11)
  * Baseline hyperleukocytosis ≥ 100 g/L or progression of leukocytosis or extra-medullary localizations despite treatment with hydroxyurea
* No AML with favorable or intermediate prognosis
* No AML secondary to myelodysplastic syndrome diagnosed within the past 3 months or myeloproliferative syndrome

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Total bilirubin < 35 μmol/L
* Transaminases < 2.5 times upper limit of normal in the absence of leukemia-related abnormalities
* Creatinine < 170 μmol/L OR creatinine clearance ≥ 50 mL/min in the absence of leukemia-related abnormalities
* Not pregnant or nursing
* Normal cardiac function by LVEF (echographic ≥ 40% or isotopic ≥ 50%)
* Affiliated with a social security system
* No uncontrolled or severe cardiovascular disease, including any of the following:

  * Myocardial infarction within the past 3 months
  * Cardiac insufficiency
  * Uncontrolled arrhythmia
* No other active cancer within the past year except for basal cell carcinoma of the skin or epithelioma in situ of the cervix
* No patients deprived of freedom or under guardianship (including temporary guardianship)
* No psychological, familial, geographical, or social situations that preclude follow-up
* No other contraindications to study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior hydroxyurea allowed
* No concurrent disulfiram
* No concurrent participation in another study with an experimental drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (phase I)
Rate of complete remission (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Vey, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France